CLINICAL TRIAL: NCT00857298
Title: Effect of Diet-induced Weight Loss on HIV-associated Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HW-08-0628
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: HIV (Human Immunodeficiency Virus); Metabolic Syndrome; HIV Infections
Keywords: HIV; Metabolic Syndrome; Obesity; Treatment Experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Metabolic Syndrome; HIV Infections; Obesity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV-MS (Active Comparator): HIV-positive obese women with metabolic syndrome will be studied before and after losing 6-8% of body weight
  Interventions: Behavioral: Dietary Intervention
- MS only (Active Comparator): HIV-negative obese women with metabolic syndrome will be studied before and after losing 6-8% of body weight
  Interventions: Behavioral: Dietary Intervention

INTERVENTIONS:
Behavioral: Dietary Intervention — The nutrition curriculum will involve weekly group and individual sessions. The initial calorie goal will be ~750 kcal below the resting energy equivalent, and adjusted as needed to achieve weight loss targets.

SUMMARY:
Obese HIV-positive women with Metabolic Syndrome (HIV-MS) and obese HIV-negative women with Metabolic Syndrome will be studied before and after achieving moderate (6%-8%) diet-induced weight loss. The investigators hypothesize that health markers will improve in both groups but that the improvement will be blunted in the women with HIV-MS.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary
* Obese
* Have either dyslipidemia (HDL < 50 or triglycerides > 150), waist circumference > 88cm, and impaired glucose tolerance or homeostasis model assessment value of > 3
* Subjects with HIV-MS must have been receiving HAART for > 6 months

Exclusion Criteria:

* Medication changes in the last 3 months
* Diabetes mellitus
* Medical problems that in the opinion of the principal investigator may interfere with patient safety
* Substance abuse

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Effect of weight loss on body composition | three months
Effect of weight loss on insulin action | three months

SECONDARY OUTCOMES:
Effect of weight loss on body fat mass | three months
Effect of weight loss on adipose tissue distribution | three months
Effect of weight loss intrahepatic triglyceride content | three months
Effect of weight loss on insulin action adipose tissue | three months
Effect of weight loss on insulin action in liver | three months
Effect of weight loss on insulin action in skeletal muscle | three months

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Reeds, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Reeds DN, Pietka TA, Yarasheski KE, Cade WT, Patterson BW, Okunade A, Abumrad NA, Klein S. HIV infection does not prevent the metabolic benefits of diet-induced weight loss in women with obesity. Obesity (Silver Spring). 2017 Apr;25(4):682-688. doi: 10.1002/oby.21793. Epub 2017 Feb 28. PMID 28245099